CLINICAL TRIAL: NCT01164501
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel Group, Efficacy and Safety Study of BI 10773 (10 mg and 25 mg Administered Once Daily) as Add on to Pre-existing Antidiabetic Therapy Over 52 Weeks in Patients With Type 2 Diabetes Mellitus and Renal Impairment and Insufficient Glycaemic Control
Brief Title: Efficacy and Safety of Empagliflozin (BI 10773) in Patients With Type 2 Diabetes and Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.36; 2009-016179-31 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — empagliflozin

ARMS (3):
- BI 10773 low dose (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- BI 10773 high dose (Experimental): BI 10773 tablets once daily
  Interventions: Drug: Placebo; Drug: BI 10773
- Placebo (Placebo Comparator): Placebo tablets matching BI 10773
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 low dose
Drug: Placebo — Placebo tablets identical to BI 10773 low dose
  Arms: BI 10773 high dose
Drug: Placebo — Placebo tablets identical to BI 10773 high dose
  Arms: Placebo
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 high dose
Drug: Placebo — Placebo tablets identical to BI 10773 low dose
  Arms: Placebo
Drug: Placebo — Placebo tablets identical to BI 10773 high dose
  Arms: BI 10773 low dose

SUMMARY:
This study will investigate the efficacy and safety of the BI 10773 in type 2 diabetic patients with renal impairment in order to provide these data for approval for BI 10773 as an antidiabetic agent by regulatory authorities.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent and an estimated glomerular filtration rate of <90 ml/min.
2. Male and female patients on diet and exercise regimen who are pre-treated with any antidiabetic therapy and are on the maximum tolerated dose which has been unchanged for 12 weeks prior to randomisation.
3. HbA1c greater than or equal to 7.0% and less than or equal to 10.0% .
4. Aged 18 years or above.
5. Body Mass Index less than or equal to 45 kg/m2

Exclusion criteria:

1. Uncontrolled hyperglycaemia defined as >13.3 mmol/L after an overnight fast during placebo run-in.
2. Impaired renal function, defined as an estimated glomerular filtration rate <15 ml/min.
3. Renal impairment requiring any form of chronic dialysis.
4. Requiring acute dialysis within three months prior to informed consent.
5. Renal transplant recipient.
6. Myocardial infarction, stroke or Transient Ischemic Attack within three months prior to informed consent.
7. Indication of liver disease.
8. Bariatric surgery within the past two years.
9. Medical history of cancer.
10. Blood dyscrasias or any disorders causing hemolysis or unstable red blood cell.
11. Contraindications to pre-existing background antidiabetic therapy.
12. Treatment with anti-obesity drugs.
13. Current treatment with systemic steroids or change in dosage of thyroid hormones within six weeks prior to informed consent or any other uncontrolled endocrine disorder except Type 2 Diabetes.
14. Pre-menopausal women who are nursing or pregnant or are of child-bearing potential and are not practising an acceptable method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (127):
- United States (18):
  - 1245.36.10014 Boehringer Ingelheim Investigational Site, Anaheim, California
  - 1245.36.10019 Boehringer Ingelheim Investigational Site, Lomita, California
  - 1245.36.10017 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 1245.36.10009 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 1245.36.10018 Boehringer Ingelheim Investigational Site, Honolulu, Hawaii
  - 1245.36.10015 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1245.36.10021 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 1245.36.10008 Boehringer Ingelheim Investigational Site, Greenville, North Carolina
  - 1245.36.10005 Boehringer Ingelheim Investigational Site, Bethlehem, Pennsylvania
  - 1245.36.10003 Boehringer Ingelheim Investigational Site, Melrose Park, Pennsylvania
  - 1245.36.10004 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1245.36.10012 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 1245.36.10013 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1245.36.10002 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1245.36.10007 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1245.36.10023 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 1245.36.10011 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1245.36.10006 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Canada (9):
  - 1245.36.20052 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1245.36.20054 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1245.36.20023 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1245.36.20055 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1245.36.20048 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1245.36.20051 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1245.36.20086 Boehringer Ingelheim Investigational Site, Thornhill, Ontario
  - 1245.36.20053 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1245.36.20056 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- France (9):
  - 1245.36.33001 Boehringer Ingelheim Investigational Site, Corbeil-Essonnes
  - 1245.36.33042 Boehringer Ingelheim Investigational Site, Nanterre
  - 1245.36.33041 Boehringer Ingelheim Investigational Site, Nice
  - 1245.36.33036 Boehringer Ingelheim Investigational Site, Paris
  - 1245.36.33040 Boehringer Ingelheim Investigational Site, Poitiers
  - 1245.36.33037 Boehringer Ingelheim Investigational Site, Reims
  - 1245.36.33038 Boehringer Ingelheim Investigational Site, Reims
  - 1245.36.33043 Boehringer Ingelheim Investigational Site, Rennes
  - 1245.36.33044 Boehringer Ingelheim Investigational Site, Saint-Mandé
- Hong Kong (5):
  - 1245.36.85201 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.36.85204 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.36.85205 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.36.85206 Boehringer Ingelheim Investigational Site, Hong Kong
  - 1245.36.85202 Boehringer Ingelheim Investigational Site, Kowloon
- India (15):
  - 1245.36.91209 Boehringer Ingelheim Investigational Site, Aligarh, Uttar Pradesh
  - 1245.36.91202 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.36.91204 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.36.91205 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.36.91208 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.36.91201 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.36.91214 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.36.91213 Boehringer Ingelheim Investigational Site, Gūrgaon
  - 1245.36.91203 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1245.36.91211 Boehringer Ingelheim Investigational Site, Kolkata
  - 1245.36.91210 Boehringer Ingelheim Investigational Site, Mangalore
  - 1245.36.91215 Boehringer Ingelheim Investigational Site, Mumbai, Maharastra
  - 1245.36.91216 Boehringer Ingelheim Investigational Site, Nashik
  - 1245.36.91212 Boehringer Ingelheim Investigational Site, New Delhi
  - 1245.36.91207 Boehringer Ingelheim Investigational Site, Pune
- Malaysia (10):
  - 1245.36.60003 Boehringer Ingelheim Investigational Site, Johor Baru
  - 1245.36.60006 Boehringer Ingelheim Investigational Site, Kelantan Kota Bahru
  - 1245.36.60005 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1245.36.60009 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1245.36.60004 Boehringer Ingelheim Investigational Site, Kuala Pahang
  - 1245.36.60007 Boehringer Ingelheim Investigational Site, Perak
  - 1245.36.60011 Boehringer Ingelheim Investigational Site, Perak
  - 1245.36.60010 Boehringer Ingelheim Investigational Site, Pulau Piang
  - 1245.36.60008 Boehringer Ingelheim Investigational Site, Sabak Bernam
  - 1245.36.60001 Boehringer Ingelheim Investigational Site, Selangor Darul Ehsan
- Netherlands (7):
  - 1245.36.31015 Boehringer Ingelheim Investigational Site, Amersfoort
  - 1245.36.31012 Boehringer Ingelheim Investigational Site, Geleen
  - 1245.36.31017 Boehringer Ingelheim Investigational Site, Hardenberg
  - 1245.36.31009 Boehringer Ingelheim Investigational Site, Maastricht
  - 1245.36.31004 Boehringer Ingelheim Investigational Site, The Hague
  - 1245.36.31002 Boehringer Ingelheim Investigational Site, Utrecht
  - 1245.36.31003 Boehringer Ingelheim Investigational Site, Zaandam
- Philippines (6):
  - 1245.36.63008 Boehringer Ingelheim Investigational Site, Cavite City
  - 1245.36.63006 Boehringer Ingelheim Investigational Site, Cebu
  - 1245.36.63005 Boehringer Ingelheim Investigational Site, Manila
  - 1245.36.63007 Boehringer Ingelheim Investigational Site, Manila
  - 1245.36.63009 Boehringer Ingelheim Investigational Site, Marikina City
  - 1245.36.63010 Boehringer Ingelheim Investigational Site, Tacloban City
- Poland (7):
  - 1245.36.48006 Boehringer Ingelheim Investigational Site, Gdansk
  - 1245.36.48003 Boehringer Ingelheim Investigational Site, Lodz
  - 1245.36.48004 Boehringer Ingelheim Investigational Site, Lodz
  - 1245.36.48001 Boehringer Ingelheim Investigational Site, Lublin
  - 1245.36.48002 Boehringer Ingelheim Investigational Site, Poznan
  - 1245.36.48007 Boehringer Ingelheim Investigational Site, Ruda Śląska
  - 1245.36.48005 Boehringer Ingelheim Investigational Site, Torun
- Portugal (4):
  - 1245.36.35003 Boehringer Ingelheim Investigational Site, Faro
  - 1245.36.35002 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.36.35004 Boehringer Ingelheim Investigational Site, Lisbon
  - 1245.36.35001 Boehringer Ingelheim Investigational Site, Vila Nova de Gaia
- Russia (6):
  - 1245.36.70008 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.36.70009 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.36.70011 Boehringer Ingelheim Investigational Site, Moscow
  - 1245.36.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.36.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1245.36.70002 Boehringer Ingelheim Investigational Site, Vsevolozhsk
- Slovakia (6):
  - 1245.36.74011 Boehringer Ingelheim Investigational Site, Moldava nad Bodvou
  - 1245.36.74013 Boehringer Ingelheim Investigational Site, Nitra
  - 1245.36.74008 Boehringer Ingelheim Investigational Site, Nové Mesto nad Váhom
  - 1245.36.74012 Boehringer Ingelheim Investigational Site, Prešov
  - 1245.36.74007 Boehringer Ingelheim Investigational Site, Trenčín
  - 1245.36.74009 Boehringer Ingelheim Investigational Site, Žilina
- South Africa (3):
  - 1245.36.76021 Boehringer Ingelheim Investigational Site, Plumstead
  - 1245.36.76020 Boehringer Ingelheim Investigational Site, Somerset West
  - 1245.36.76022 Boehringer Ingelheim Investigational Site, Somerset West
- Spain (10):
  - 1245.36.34015 Boehringer Ingelheim Investigational Site, Barcelona
  - 1245.36.34009 Boehringer Ingelheim Investigational Site, Granada
  - 1245.36.34014 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1245.36.34012 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.36.34013 Boehringer Ingelheim Investigational Site, Madrid
  - 1245.36.34020 Boehringer Ingelheim Investigational Site, Manresa
  - 1245.36.34021 Boehringer Ingelheim Investigational Site, San Sebastián de los Reyes
  - 1245.36.34016 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 1245.36.34017 Boehringer Ingelheim Investigational Site, Valencia
  - 1245.36.34019 Boehringer Ingelheim Investigational Site, Valencia
- United Kingdom (12):
  - 1245.36.44018 Boehringer Ingelheim Investigational Site, Bath
  - 1245.36.44010 Boehringer Ingelheim Investigational Site, Birmingham
  - 1245.36.44013 Boehringer Ingelheim Investigational Site, Blackpool
  - 1245.36.44016 Boehringer Ingelheim Investigational Site, Blackpool
  - 1245.36.44026 Boehringer Ingelheim Investigational Site, Chester
  - 1245.36.44012 Boehringer Ingelheim Investigational Site, Chesterfield
  - 1245.36.44025 Boehringer Ingelheim Investigational Site, Doncaster
  - 1245.36.44036 Boehringer Ingelheim Investigational Site, Epsom
  - 1245.36.44001 Boehringer Ingelheim Investigational Site, Frome
  - 1245.36.44007 Boehringer Ingelheim Investigational Site, Midsomer Norton
  - 1245.36.44023 Boehringer Ingelheim Investigational Site, Nantwich
  - 1245.36.44024 Boehringer Ingelheim Investigational Site, Welwyn Garden City

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Cherney D, Lund SS, Perkins BA, Groop PH, Cooper ME, Kaspers S, Pfarr E, Woerle HJ, von Eynatten M. The effect of sodium glucose cotransporter 2 inhibition with empagliflozin on microalbuminuria and macroalbuminuria in patients with type 2 diabetes. Diabetologia. 2016 Sep;59(9):1860-70. doi: 10.1007/s00125-016-4008-2. Epub 2016 Jun 17. PMID 27316632
- [Derived] Barnett AH, Mithal A, Manassie J, Jones R, Rattunde H, Woerle HJ, Broedl UC; EMPA-REG RENAL trial investigators. Efficacy and safety of empagliflozin added to existing antidiabetes treatment in patients with type 2 diabetes and chronic kidney disease: a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2014 May;2(5):369-84. doi: 10.1016/S2213-8587(13)70208-0. Epub 2014 Jan 24. PMID 24795251

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablets, matching the empagliflozin 10mg and 25mg tablets, taken once daily for 52 weeks.
- Empa 10mg: Single oral dose of empagliflozin (empa) 10mg plus a placebo tablet matching the 25mg empa dose were taken once daily for 52 weeks.
- Empa 25mg: Single oral dose of empagliflozin (empa) 25mg plus a placebo tablet matching the 10mg empa dose were taken once daily for 52 weeks.
Period: Overall Study
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Started | 321 | 98 | 322
Completed | 278 | 88 | 280
Not Completed | 43 | 10 | 42
Not completed — Not treated | 2 | 0 | 1
Not completed — Adverse Event | 18 | 4 | 21
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Non compliant with protocol | 1 | 1 | 4
Not completed — Lost to Follow-up | 3 | 0 | 3
Not completed — Patient refusal to continue,not due toAE | 10 | 4 | 8
Not completed — Other reason not defined above | 9 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for treated patients only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empa 10mg | Empa 25mg | Total
Number analyzed (Participants) | 319 | 98 | 321 | 738
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.7) | 63.2 (8.5) | 63.9 (9.0) | 63.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 38 | 132 | 308
  Male | 181 | 60 | 189 | 430

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline in Patients With Mild or Moderate Renal Impairment
Description: Change from baseline in HbA1c after 24 weeks, for patients with mild or moderate renal impairment.
  Note adjusted means are provided.
Time Frame: Baseline and 24 weeks
Population: Full analysis set (FAS) which included all randomised patients, treated with at least one dose of trial medication, who had a baseline HbA1c value. Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empa 25mg
Number analyzed (Participants) | 282 | 284
percentage of HbA1c | 0.05 (0.04) | -0.46 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons, no adjustment in p-values. Empa 25 mg versus placebo in mild or moderate renal impaired patients was the first step in the hierarchical sequence; Based on ANCOVA with terms for treatment, background antidiabetic medication, renal impairment and baseline HbA1c; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.62 to -0.39], Standard Error of Mean 0.06 — Difference calculated as empa 25mg minus placebo

2. Primary Outcome: HbA1c Change From Baseline in Patients With Mild Renal Impairment
Description: Change from baseline in HbA1c after 24 weeks, for patients with mild renal impairment.
  Note adjusted means are provided.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 95 | 98 | 97
percentage of HbA1c | 0.06 (0.07) | -0.46 (0.07) | -0.63 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons, no adjustment in p-values. Empa 25 mg versus placebo in mild renal impaired patients was the second step in the hierarchical sequence; Based on ANCOVA with terms for treatment, background antidiabetic medication and baseline HbA1c; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.72 to -0.32], Standard Error of Mean 0.10 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons, no adjustment in p-values. Empa 10 mg versus placebo in mild renal impaired patients was the third step in the hierarchical sequence; Based on ANCOVA with terms for treatment, background antidiabetic medication and baseline HbA1c; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-0.88 to -0.49], Standard Error of Mean 0.10 — Difference calculated as empa 25mg minus placebo

3. Primary Outcome: HbA1c Change From Baseline in Patients With Moderate Renal Impairment
Description: Change from baseline in HbA1c after 24 weeks, for patients with moderate renal impairment.
  Note adjusted means are provided.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Placebo: Placebo tablet, matching the empagliflozin 10mg and 25mg tablets, taken once daily for 52 weeks.
Arm/Group | Placebo | Empa 25mg
Number analyzed (Participants) | 187 | 187
percentage of HbA1c | 0.05 (0.05) | -0.37 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons, no adjustment in p-values. Empa 10 mg versus placebo in moderate renal impaired patients was the fourth step in the hierarchical sequence; Based on ANCOVA with terms for treatment, background antidiabetic medication and baseline HbA1c; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.56 to -0.28], Standard Error of Mean 0.07 — Difference calculated as empa 25mg minus placebo

4. Other Pre Specified Outcome: Hypoglycaemic Events
Description: Percentage of patients who experienced a hypoglycaemic event. A hypoglycaemic event was regarded as confirmed if it was documented as an adverse event with plasma glucose values <= 70 mg/dL (<=3.9mmol/L) measured or with a documentation that the assistance of another person to actively administer carbohydrate, glucagon or other resuscitative action had been required.
Time Frame: From first drug administration until 7 days after last trial medication intake, up to 458 days
Population: Treated set which included all patients treated with at least one dose of randomised trial medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 319 | 98 | 321
percentage of participants | 27.6 | 26.5 | 27.4

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after last trial medication intake, up to 458 days
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Serious Adverse Events (participants affected / at risk) | 44/319 | 6/98 | 40/321
Other Adverse Events (participants affected / at risk) | 207/319 | 64/98 | 187/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=319) | Empa 10mg (N=98) | Empa 25mg (N=321)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 3 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2
Dengue fever (Infections and infestations) | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 3
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 0 | 3
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Intra-abdominal haematoma (Vascular disorders) | 1 | 0 | 0
Lymphocele (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=319) | Empa 10mg (N=98) | Empa 25mg (N=321)
Balanitis candida (Infections and infestations) | 0 | 5 | 0
Influenza (Infections and infestations) | 8 | 6 | 8
Nasopharyngitis (Infections and infestations) | 29 | 6 | 27
Upper respiratory tract infection (Infections and infestations) | 25 | 14 | 35
Urinary tract infection (Infections and infestations) | 39 | 14 | 38
Hyperglycaemia (Metabolism and nutrition disorders) | 41 | 4 | 23
Hypoglycaemia (Metabolism and nutrition disorders) | 92 | 27 | 89
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 7 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 8 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 8 | 6
Headache (Nervous system disorders) | 13 | 5 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 2 | 11
Hypertension (Vascular disorders) | 20 | 1 | 14

LIMITATIONS AND CAVEATS:
In this trial, only patients with mild or moderate renal impairment were analysed. Patients with severe or no renal impairment were not analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.